CLINICAL TRIAL: NCT06424431
Title: Stapler Versus Stapler Combined With Electrocautery for Pancreatic Transection and Stump Closure for Distal Pancreatectomy
Brief Title: Methods of Pancreatic Stump Closure for Distal Pancreatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2024-110
Record Dates: First submitted 2024-04-03; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Pancreatectomy
MeSH Terms: interventions — Electrocoagulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stapler (Other): Simple closure with a closure device for closure of the pancreatic remnant in distal pancreatectomy.
  Interventions: Procedure: simple closure with a closure device
- Stapler combined with electrocautery (Experimental): Closure with a closure device combined with electrocoagulation for closure of the pancreatic remnant in distal pancreatectomy.
  Interventions: Procedure: stapler combined with electrocautery

INTERVENTIONS:
Procedure: stapler combined with electrocautery — Closure with a closure device combined with electrocoagulation for pancreatic stump closure in distal pancreatectomy
  Arms: Stapler combined with electrocautery
Procedure: simple closure with a closure device — Simple closure with a closure device for pancreatic stump closure in distal pancreatectomy
  Arms: Stapler

SUMMARY:
The aim of this study is to conduct a retrospective analysis of patients who underwent distal pancreatectomy in our hospital, aiming to evaluate the safety and feasibility of two methods for closure of the pancreatic remnant: simple closure with a closure device and closure combined with electrocoagulation.

DETAILED DESCRIPTION:
The aim of this study is to conduct a retrospective analysis of patients who underwent distal pancreatectomy in our hospital, aiming to evaluate the safety and feasibility of two methods for closure of the pancreatic remnant: simple closure with a closure device and closure combined with electrocoagulation. This study aims to determine which method is safer and more feasible, with the potential to reduce postoperative complications, improve outcomes, facilitate better patient recovery, and thereby provide better guidance for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent distal pancreatectomy performed by Director Jin Gang's team at Changhai Hospital affiliated with Naval Medical University between January 2019 and January 2023.
* Patients who underwent closure of the pancreatic remnant using either simple closure or closure combined with electrocoagulation during surgery.

Exclusion Criteria:

* Patients undergoing surgeries by other primary clinical teams during the same period.
* Patients undergoing closure of the pancreatic remnant using methods other than those mentioned.
* Patients who violate the requirements of the study protocol.
* Patients with incomplete data collection in the hospital's diagnostic and treatment system.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula | perioperatively
  Postoperative pancreatic fistula

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China